CLINICAL TRIAL: NCT01943968
Title: Lysyl Oxidase, Semaphorin 7a and Semaphorin 3a in Patients With Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-075-13
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Systemic sclerosis patients (Other): Systemic sclerosis patients will have blood tested for fibrotic enzyme levels
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test

SUMMARY:
The aim of our study is to find a biomarker for fibrosis or vasculopathy in systemic sclerosis. We will evaluate a possible correlation between semaphorin 7a, semaphorin 3a and lysyl oxidase and fibrosis (lung and skin) or vasculopathy in patients with systemic sclerosis. The results obtained may help us diagnose these complications of systemic sclerosis and hopefully even monitor patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Sclerosis Patients
* Written consent to participation in study

Exclusion Criteria:

* Serious active medical condition
* Other autoimmune rheumatic disease
* Current or past allergic/inflammatory reaction
* Liver disease
* Pregnant or breastfeeding
* Illegal drug or alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Fibrin Enzyme Levels in Blood | Six months
  Patients will undergo blood tests before study and after six months to determine levels of lysyl oxidase, semaphorin 7a and 3a and thus determine severity of the disease (systemic sclerosis).

CONTACTS AND LOCATIONS:
Overall Officials: Doron River, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel